CLINICAL TRIAL: NCT05938387
Title: A Phase 1 Dose-Finding Study to Evaluate Safety and Tolerability of CVGBM in Patients with Surgically Resected Glioblastoma (GBM) or Astrocytoma with a Molecular Signature of Unmethylated Glioblastoma
Brief Title: Safety and Tolerability of CVGBM in Adults with Newly Diagnosed MGMT-Unmethylated Glioblastoma or Astrocytoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: CureVac (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CV-GBLM-001; 2022-501423-25 (EudraCT Number)
Record Dates: First submitted 2023-06-06; First posted 2023-07-10 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Dose escalation: CVGBM Dose Level -1 (Experimental): Dose Level -1 represents a dose that may be evaluated if dose level 1 is poorly tolerated. No dose de-escalation below this level is planned for this study. If the dose level -1 is poorly tolerated, the study will be terminated.
  Interventions: Biological: CV09050101 mRNA vaccine (CVGBM) 6 μg
- Dose escalation: CVGBM Dose Level 1 (Experimental)
  Interventions: Biological: CV09050101 mRNA vaccine (CVGBM) 12 μg
- Dose escalation: CVGBM Dose Level 2 (Experimental)
  Interventions: Biological: CV09050101 mRNA vaccine (CVGBM) 25 μg
- Dose escalation: CVGBM Dose Level 3 (Experimental)
  Interventions: Biological: CV09050101 mRNA vaccine (CVGBM) 50 μg
- Dose escalation: CVGBM Dose Level 4 (Experimental)
  Interventions: Biological: CV09050101 mRNA vaccine (CVGBM) 100 μg
- Dose expansion (Experimental): After completion of the dose-escalation part and safety data review by the DSMB, approximately 20 patients will be enrolled at the selected Recommended Dose for Expansion (RDE) to generate more data on safety, tolerability and immunogenicity.
  Interventions: Biological: CV09050101 mRNA vaccine RDE 100 μg

INTERVENTIONS:
Biological: CV09050101 mRNA vaccine (CVGBM) 12 μg — CVGBM will be administered as an IM injection.
  Arms: Dose escalation: CVGBM Dose Level 1
Biological: CV09050101 mRNA vaccine (CVGBM) 25 μg — CVGBM will be administered as an IM injection.
  Arms: Dose escalation: CVGBM Dose Level 2
Biological: CV09050101 mRNA vaccine (CVGBM) 50 μg — CVGBM will be administered as an IM injection.
  Arms: Dose escalation: CVGBM Dose Level 3
Biological: CV09050101 mRNA vaccine (CVGBM) 100 μg — CVGBM will be administered as an IM injection.
  Arms: Dose escalation: CVGBM Dose Level 4
Biological: CV09050101 mRNA vaccine RDE 100 μg — CVGBM will be administered as an IM injection.
  Arms: Dose expansion
Biological: CV09050101 mRNA vaccine (CVGBM) 6 μg — CVGBM will be administered as an IM injection.
  Arms: Dose escalation: CVGBM Dose Level -1

SUMMARY:
This study is an open-label, first-in-human, dose-escalation study of CV09050101 mRNA vaccine (CVGBM) in patients with newly diagnosed "MGMT-unmethylated" Glioblastoma (GBM). Patients with isocitrate dehydrogenase (IDH)-wildtype astrocytoma with a molecular signature of "unmethylated" GBM are also eligible.

After surgical resection and completion of radiotherapy for GBM with or without chemotherapy, patients will receive CVGBM i.e. as monotherapy after radiotherapy with or without chemotherapy.

The study consists of a dose-escalation part (Part A) which completes enrollment in February 2024 and a dose-expansion part (Part B) which is anticipated to begin enrolling in June/July 2024.

Patients will receive a total of 7 administrations of CVGBM on Days 1, 8, 15, 29, 43, 57, and 71. At the discretion of the Investigator in alignment with the Sponsor's medical monitor the vaccinations may continue beyond Day 71 every 6 weeks until one year after the first CVGBM vaccination or upon disease progression or undue toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed, newly diagnosed GBM (CNS WHO Grade 4) and IDH-wildtype astrocytoma with a molecular signature of "unmethylated" GBM.
2. Specific HLA genotype.
3. Gross total or partial resection (i.e., ≥50% of tumor volume resected).
4. Having completed radiotherapy with or without chemotherapy post-surgery at least 2 weeks before study treatment initiation with no signs of disease progression. Patients must have recovered from any radiotherapy or chemotherapy related side effects to ≤ Grade 1 (with the exception of ALC and WBC as per eligibility criteria). Pretreatment (and concomitant treatment) with TTFields therapy for GBM is allowed.
5. Age ≥18 years.
6. Karnofsky Performance Status (KPS) ≥70%.
7. Life expectancy >6 months.
8. Absolute lymphocyte count (ALC) >0.5 x109/L.
9. Each patient must voluntarily sign and date an informed consent form (ICF) approved by an Independent Ethics Committee (IEC), prior to the initiation of any pre-screening, screening or study-specific procedures. Note: Patients will sign a separate ICF to allow pre-screening/HLA genotyping.
10. Female patients who are post-menopausal (no menses for at least 12 months before the Screening Visit), or surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy).

    Females of childbearing potential must:
    1. Have a negative serum pregnancy test with a sensitivity of at least 25 mIU/mL within 10 to 14 days, and within 24 hours prior to starting the study treatment a negative urine pregnancy test.
    2. Agree to ongoing pregnancy testing during the study.
    3. Use effective contraception at least 28 days before starting study treatment through to 30 days after the last dose of study treatment. Effective methods of birth control include:

       * combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation:

         * oral
         * intravaginal
         * transdermal
       * progestogen-only hormonal contraception associated with inhibition of ovulation:

         * oral
         * injectable
         * implantable
       * intrauterine device
       * intrauterine hormone-releasing system
       * bilateral tubal occlusion
       * vasectomised partner + barrier method
       * sexual abstinence: Either agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal (coitus interruptus), spermicides only and lactational amenorrhoea method (LAM) are not acceptable methods of contraception.
11. Male patients, even if surgically sterilized (i.e., status postvasectomy), must:

    1. Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal (coitus interruptus), spermicides only and LAM are not acceptable methods of contraception.
    2. Agree to practice effective barrier contraception during the entire study treatment period (e.g., condom) and through to 3 months after the last dose of study treatment if their partner is of childbearing potential, even if they have had a successful vasectomy.

Exclusion Criteria:

1. Abnormal (≥Grade 2 NCI-CTCAE v5.0) laboratory values for hematology, liver and renal function (serum creatinine). The following values apply as exclusion criteria:

   1. Hemoglobin <10 g/dL (6.2 mmol/L)
   2. White blood cell (WBC) count decrease (<2.5 x109/L)
   3. Absolute neutrophil count (ANC) decrease <1.5 x109/L
   4. Platelet count decrease <75 x109/L
   5. Bilirubin >1.5 x upper limit of normal (ULN according to the performing lab's reference range), except for patients with Gilbert's syndrome
   6. Alanine aminotransferase (ALT) >3 x ULN
   7. Aspartate aminotransferase (AST) >3 x ULN
   8. Gamma glutamyltransferase (GGT) >2.5 x ULN
   9. Serum creatinine increased >1.5 x ULN
2. Tumor biopsy only without gross total or partial resection (i.e., ≥50% of tumor volume resected).
3. Any prior therapy for GBM (except surgery, radiotherapy with or without chemotherapy (e.g., temozolomide [TMZ]), TTFields, and steroids) including immunotherapy.
4. Patient on stable or decreasing steroid levels exceeding 10 mg/day prednisone (or equivalent doses of other steroids) during the last 3 days prior to enrollment. Expectation that the patient will need steroid doses >10 mg/day prednisone or equivalent during the next 3 months. Note: Steroid treatment during the study will be allowed for treatment of cerebral edema or other life-threatening conditions.
5. Active human immunodeficiency virus (HIV) infection (ie, CD4 count below the normal range) or active Hepatitis B or C infection (i.e., detectable levels of Hepatitis B DNA or Hepatitis C RNA), or active infections requiring oral or intravenous antibiotics or that can cause a severe disease.
6. Clinically relevant autoimmune diseases that could impact the assessment of vaccine safety and efficacy (with the exception of clinically stable thyroid diseases under medication and vitiligo).
7. Immunosuppression, not related to prior treatment for malignancy. Any medical condition that requires chronic systemic immunosuppressive therapy including chronic corticosteroids (except physiologic maintenance/replacement doses), methotrexate, tacrolimus or any other immunosuppressive agents within 28 days of treatment start, including, but not limited, to organ transplant-related immunosuppression.
8. Patients with prior hematopoietic stem cell transplantation/prior organ allograft.
9. Any condition that in the judgment of the Investigator is likely to prevent compliance with study procedures.
10. Patients with impaired coagulation or any bleeding disorder in whom an intramuscular injection or blood draw is contraindicated.
11. History of myocarditis or pericarditis within the last 3 months or history of myocarditis or pericarditis following COVID-19 vaccination.
12. Previous mRNA vaccination (e.g., SARS-CoV2) or live attenuated vaccination within 1 month prior to study treatment initiation, other vaccines within 2 weeks prior to study treatment initiation.
13. Serious illness or condition, which according to the Investigator poses an undue risk for the patient when participating in the trial, including, but not limited to, any of the following:

    1. Clinically significant cardiovascular disease (myocardial infarction or stroke within last 6 months, uncontrolled angina within last 3 months, diagnosed or suspected clinically significant ventricular arrhythmias, ejection fraction <35%, cerebrovascular event within last 6 months, uncontrolled hypertension [blood pressure ≥180 mm Hg systolic and 110 mmHg diastolic despite medication])
    2. New York Heart Association Class III to IV congestive heart failure
    3. Symptomatic peripheral vascular disease
    4. Severe pulmonary disease (e.g., severe chronic obstructive pulmonary disease, pneumonitis or interstitial lung disease)
    5. Uncontrolled diabetes (repeated episodes of severe hypo- or hyperglycemia requiring hospitalization)
    6. Severe mental retardation/impairment, psychiatric conditions or substance abuse resulting in inability to understand informed consent or affecting the patient's cooperation in the study
    7. Severe infection/inflammatory conditions
14. History of other malignancies (except for those which have been adequately treated and have had no recurrence).
15. Previous anaphylactic or severe allergic reaction to an LNP formulated drug or vaccine (e.g., Comirnaty or Spikevax) or known allergy to any other component of CVGBM (e.g., PEG).
16. Allergy to aminoglycoside antibiotics.
17. Pregnant or breastfeeding.
18. Prior (within 30 days prior to study enrollment) or concurrent participation in another interventional clinical trial studying an investigational product, drug or treatment regimen. At least 30 days should have passed prior to the first study treatment with the investigational product (exceptions may be considered on a case-by-case basis after consultation with the CureVac Medical Director).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-02-04 (Estimated); Study Completion 2026-02-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-related adverse events (TRAEs) | 1 year
Incidence of treatment-emergent adverse events (TEAEs) | 1 year
Incidence of serious adverse events (SAEs) | 1 year
Incidence of immune related adverse events (irAEs) | 1 year
Incidence of injection site reactions (ISRs) | 1 year
Incidence of clinically significant laboratory abnormalities per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v.5.0 | 1 year
Incidence dose-limiting toxicities (DLTs) | Through the first 2 weeks of treatment
Severity of DLTs (Unit: Grading via NCI-CTCAE v5.0) | Through the first 2 weeks of treatment

SECONDARY OUTCOMES:
Time to relapse from the day of surgery until the last scheduled visit of the study | 1 year
Progression-Free Survival (PFS) rate from the day of surgery until the last scheduled visit of the study | 1 year
Overall survival (OS) rate from the day of surgery until the last scheduled visit of the study | 1 year
Change in the patients' quality of life measured using a patient-reported-outcome questionnaire | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Information, Study Director — CureVac SE
Locations (13):
- Belgium (2):
  - Universitair Ziekenhuis Brussel - PPDS, Brussels
  - CHU de Liège, Liège
- Germany (10):
  - Universitätsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - University Clinic Heidelberg, Heidelberg, Baden-Wurttemberg
  - Universitätsmedizin Mannheim, Mannheim, Baden-Wurttemberg
  - Universitätsklinikum Tübingen, Tübingen, Baden-Wurttemberg
  - University Clinic Regensburg, Regensburg, Bavaria
  - Universitätsklinikum Frankfurt, Frankfurt am Main, Hesse
  - Universitätsklinikum Bonn, Bonn, North Rhine-Westphalia
  - University Hospital Essen, Essen, North Rhine-Westphalia
  - Universitatsklinikum Leipzig, Leipzig, Saxony
  - Neurosurgical Clinic at the LMU Munich, München
- Erasmusmc Cancer institute, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lutz J, Feist RK, Sonntag T, Peguero-Sanchez E, Wolter K, Bick R, Bauer J, Walz JS, Heidenreich R. Preclinical development of an mRNA-based multiepitope immunotherapeutic for glioblastoma. Cancer Immunol Immunother. 2025 Oct 6;74(11):329. doi: 10.1007/s00262-025-04178-x. PMID 41051649